CLINICAL TRIAL: NCT04351386
Title: Validation Study of the Watch HWA09 and Its Softwares ECG-SW1 and PPG-SW1 for the Detection of Atrial Fibrillation
Acronym: WEFA
Status: Completed | Type: Observational
Sponsor: Withings (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A01476-51
Record Dates: First submitted 2020-04-08; First posted 2020-04-17 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Atrial Fibrillation; Arrythmia, Cardiac
Keywords: Atrial Fibrillation; Arrythmia, Cardiac; Cardiovascular Disease; Heart Disease; Wearable Electronic Device; Watch; Electrocardiography; ECG; Photoplethysmography; PPG
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atrial Fibrillation (AF): Patients diagnosed with AF during reference ECG
  Interventions: Device: AF Detection
- Normal Sinus Rhythm (NSR): Patients with NSR during reference ECG
  Interventions: Device: AF Detection
- Other Arrythmia: Patients diagnosed with an arrhythmia other than AF during the reference ECG
  Interventions: Device: AF Detection

INTERVENTIONS:
Device: AF Detection — Recording PPG and single-lead ECG signals with the Withings HWA09 and ECG signal for the reference 12-lead ECG

SUMMARY:
The proposed clinical study aims to validate the diagnostic performance, compared to a reference ECG, of the ECG-SW1 software and the PPG-SW1 software integrated into the HWA09 watch developed by Withings for the automatic identification of atrial fibrillation (AF).

DETAILED DESCRIPTION:
HWA09 is a wrist-worn watch that enables to record a single-lead ECG similar to the standard lead I configuration, and a photoplethysmogram (PPG).

Primary objective :

To validate the diagnostic performance of the ECG-SW1 software integrated into the HWA09 watch for the automatic identification of atrial fibrillation (AF) compared to a simultaneous 12-lead ECG (hereinafter referred to as the "gold standard" or "reference method").

The algorithm classifies the watch signals into four categories: normal sinus rhythm (RSN), AF, arrhythmia other than AF, or non-interpretable. The latter category includes signals of insufficient quality to be interpreted with confidence.

This classification will be compared to the diagnosis made by three independent, blinded cardiologists based on a 12-lead ECG. The final diagnosis retained will be decided by majority with adjudication by a consensus of 3 to 6 cardiologists. The sensitivity and specificity of the device will then be estimated.

First secondary objectives:

The first secondary objective is to validate the diagnostic performance, compared to a simultaneous 12-lead ECG, of the PPG-SW1 software integrated in the HWA09 watch for the automatic identification of atrial fibrillation (AF) from the photoplethysmography (PPG) signal.

Three independent blinded cardiologists will issue a diagnosis based on the ECG recording of the HWA09 watch. The final diagnosis retained will be decided by majority with adjudication by a consensus of 3 to 6 cardiologists. Sensitivity and specificity will be calculated in relation to the reference ECG.

Second secondary objective:

To evaluate the quality of the single-channel strips measured with the HWA09 watch, as follows:

* Three independent cardiologists, having neither performed the data collection nor read the reference ECG, will independently make a diagnosis based on the HWA09 single-channel strips, blinded to the diagnosis made from the reference ECG. The ECG traces from the watch will be exported in PDF format from the Withings Health Mate application and the final diagnosis will be made by majority with adjudication by a consensus of 3 to 6 cardiologists. The final diagnosis will be compared to the diagnosis made by the cardiologists who read the reference ECG. Sensitivity and specificity will then be calculated.
* The visibility and polarity of ECG waves (i.e. P waves, QRS complex and T waves) will be determined by cardiologists for the single-channel strips recorded with HWA09 and for the lead I of the reference 12-lead ECG. For each of the waves, the agreement on their visibility and polarity (if visible) between the HWA09 and the reference ECG will be calculated.
* The durations of the major intervals of an ECG (i.e., QT interval, QRS complex, and PR interval) will be determined by the cardiologists for the single-channel strips recorded with HWA09 and for the lead I of the reference 12-lead ECG. For each interval (QT, QRS, PR), the difference of duration between the signals from the watch and the reference ECG will be calculated.
* The heart rate will first be determined by cardiologists from each signal of lead I (recorded by the HWA09 watch and the reference ECG) that has been diagnosed as NSR. The difference between the heart rate of the watch and the reference will be calculated. In a second step, the heart rate recorded by the HWA09 watch will be calculated by the Withings software. The difference between the heart rate calculated by the Withings software (from the signal of the watch) and the heart rate determined by the cardiologists (from the lead I of the reference ECG) will also be calculated.

The sponsor will ensure that no cardiologist makes a diagnosis on both a signal from the HWA09 watch and the reference ECG fomr the same patient. The sponsor will centralize diagnostics on the HWA09 and reference ECG signals and perform agreement calculations on the associated pairs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18yo
* Individuals who expressed their non-opposition to take part in the study
* Individuals affiliated to a social security system or eligible

Exclusion Criteria:

* Vulnerable individuals according to the regulation in force :

  * Pregnant, parturient or breastfeeding women
  * Individuals deprived of liberty by a court, medical or administrative order
  * Individuals under 18yo
  * Individuals legally protected or unable to express their non-opposition to take part in
  * Individuals unaffiliated to or not beneficiary of a social security system
  * Individuals who fit in multiple categories above
* Individuals having refused to take part in the study
* Individuals linguistically or mentally unable to express their non-opposition
* Individuals physically unable to wear a watch
* Individuals with an electrical pacing by a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every eligible patient doing a medical examination at the investigation center will be asked to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the automatic classification in AF by ECG-SW1 of HWA09 single-lead ECG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'
Sensitivity of the automatic classification in NSR by ECG-SW1 of HWA09 single-lead ECG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix NSR vs 'non-NSR'

SECONDARY OUTCOMES:
Sensitivity of the automatic classification in AF by PPG-SW1 of the HWA09 PPG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'
Sensitivity of the automatic classification in NSR by PPG-SW1 of the HWA09 PPG against reference 12-lead ECG | 1 year
  sensitivity from the 2x2 confusion matrix NSR vs 'non-NSR'
Sensitivity of the cardiologists' classification in AF from the HWA09 ECG | 1 year
  sensitivity from the 2x2 confusion matrix AF vs 'non-AF'
Sensitivity of the cardiologists' classification in SR from the HWA09 ECG | 1 year
  sensitivity from the 2x2 confusion matrix NSR vs 'non-NSR'
Accuracy of the visibility of P-waves of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of P-waves of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the visibility of QRS-complexes of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of QRS-complexes of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the visibility of T-waves of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
Accuracy of the positivity of T-waves of single-lead ECG from HWA09 | 1 year
  (true positives + true negatives)/(sample size) from the 2x2 confusion matrix
RMSE between cardiologist's estimate of heart rate from the HWA09 single-lead ECG and the lead I reference ECG | 1 year
  Root Mean Squared Error
RMSE between cardiologist's estimate of heart rate from the HWA09 single-lead ECG and the heart rate calculated by ECG-SW1 | 1 year
  Root Mean Squared Error

CONTACTS AND LOCATIONS:
Overall Officials: David CAMPO, Study Director — Withings; Julien NAHUM, Principal Investigator — Centre Cardiologique du Nord
Locations (3):
- France (3):
  - Institut Cœur Paris Centre Turin, Paris, Île-de-France Region
  - Hopital Europeen Georges Pompidou, Paris, Île-de-France Region
  - Centre Cardiologique du Nord, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No
Individual patient data (IPD) are considered as confidential in this study. After the end the final quality control, the database will be frozen and all the IPD will be archived .

REFERENCES:
- [Derived] Campo D, Elie V, de Gallard T, Bartet P, Morichau-Beauchant T, Genain N, Fayol A, Fouassier D, Pasteur-Rousseau A, Puymirat E, Nahum J. Atrial Fibrillation Detection With an Analog Smartwatch: Prospective Clinical Study and Algorithm Validation. JMIR Form Res. 2022 Nov 4;6(11):e37280. doi: 10.2196/37280. PMID 35481559